CLINICAL TRIAL: NCT01600079
Title: Post-Licensure Observational Study of the Long-term Effectiveness of ZOSTAVAX™
Brief Title: ZOSTAVAX™ (Zoster Vaccine Live) Long-term Effectiveness Study (V211-024)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: V211-024; 8003.016 (Other: Merck)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Herpes Zoster; Shingles
Keywords: Varicella-zoster vaccine; herpes zoster; shingles; Varicella-zoster virus; postherpetic neuralgia; Herpesviridae Infections; DNA Virus Infections; Virus Diseases
MeSH Terms: conditions — Herpes Zoster; Chickenpox; Neuralgia, Postherpetic; Herpesviridae Infections; DNA Virus Infections; Virus Diseases | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Vaccinated Cohort: Participants vaccinated with at least one dose of ZOSTAVAX™
  Interventions: Biological: ZOSTAVAX™
- Unvaccinated Comparison Cohort: Participants who are not yet vaccinated with any zoster vaccine

INTERVENTIONS:
Biological: ZOSTAVAX™ — ZOSTAVAX™ (Zoster Vaccine Live) administered in routine clinical conditions of use
  Other Names: Zoster Vaccine Live
  Groups: Vaccinated Cohort

SUMMARY:
This study will describe the impact of vaccination with ZOSTAVAX™ on the epidemiology of herpes zoster (HZ) in a cohort of vaccinated participants 50 years or age or older, compared to a cohort of unvaccinated participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with continuous Kaiser Permanente Northern California (KPNC) membership since becoming age-eligible for ZOSTAVAX™ and with 12 months of continuous enrollment in KPNC before their study start date

Exclusion Criteria:

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of Kaiser Permanente Northern California (KPNC)
Sampling Method: Non-Probability Sample
Enrollment: 1505647 (Actual)
Dates: Start 2012-05-15 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Herpes Zoster in Vaccinated and Unvaccinated Cohorts, Overall, and by Age (50-59, 60-69, 70-79 ≥80) at Vaccination | 10 years
Incidence of Herpes Zoster in Vaccinated and Unvaccinated Cohorts by Time since Vaccination | 10 years

SECONDARY OUTCOMES:
Incidence of Postherpetic Neuralgia in Vaccinated and Unvaccinated Cohorts, Overall, and by Age (50-59, 60-69, 70-79, ≥80) at Vaccination | 10 years
Incidence of Postherpetic Neuralgia in Vaccinated and Unvaccinated Cohorts by Time since Vaccination | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klein NP, Bartlett J, Fireman B, Marks MA, Hansen J, Lewis E, Aukes L, Saddier P. Effectiveness of the live zoster vaccine during the 10 years following vaccination: real world cohort study using electronic health records. BMJ. 2023 Nov 8;383:e076321. doi: 10.1136/bmj-2023-076321. PMID 37940142
- [Derived] Klein NP, Bartlett J, Fireman B, Marks MA, Hansen J, Lewis E, Aukes L, Saddier P. Long-term effectiveness of zoster vaccine live for postherpetic neuralgia prevention. Vaccine. 2019 Aug 23;37(36):5422-5427. doi: 10.1016/j.vaccine.2019.07.004. Epub 2019 Jul 10. PMID 31301920
- [Derived] Baxter R, Bartlett J, Fireman B, Marks M, Hansen J, Lewis E, Aukes L, Chen Y, Klein NP, Saddier P. Long-Term Effectiveness of the Live Zoster Vaccine in Preventing Shingles: A Cohort Study. Am J Epidemiol. 2018 Jan 1;187(1):161-169. doi: 10.1093/aje/kwx245. PMID 29309521